CLINICAL TRIAL: NCT01764568
Title: Functional Brain Networks Underlying Non-pharmaceutical Interventions for Psychosis.
Brief Title: Contrasting Group Therapy Methods for Psychosis
Acronym: MCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The full sample could not be collected due to loss of funds to complete the imaging component.
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other); Vancouver General Hospital (Other); Vancouver Coastal Health (Other Government); VGH and UBC Hospital Foundation (Other)
Responsible Party: Principal Investigator, Todd Woodward, Professor, University of British Columbia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: H12-01968; F11-02233 (Other Grant/Funding Number: Mind Foundation of British Columbia)
Record Dates: First submitted 2012-11-28; First posted 2013-01-09 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Psychosis; Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: Metacognitive training; Cognitive behavioral therapy; Clinical trial; Group intervention; Group therapy; Schizophrenia; Psychosis; Cognitive remediation
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metacognitive Training for Psychosis (Experimental): Individuals with psychosis (Schizophrenia, Schizoaffective, Schizophreniform, etc.) who will receive Metacognitive Training twice weekly for 8 weeks (16 sessions).
  Interventions: Behavioral: Metacognitive Training (MCT)
- Cognitive Remediation for Psychosis (Experimental): Individuals with psychosis (Schizophrenia, Schizoaffective, Schizophreniform, etc.) who will receive Cognitive Remediation treatment twice weekly for 8 weeks (16 sessions).
  Interventions: Behavioral: Cognitive Remediation (CR)
- Treatment as Usual for Psychosis (No Intervention): Individuals with psychosis (Schizophrenia, Schizoaffective, Schizophreniform, etc.) who will continue to receive treatment as usual (TAU) as defined by their health care team (i.e., medication, other therapies) while still taking part in baseline, midpoint, and end-point assessments.

INTERVENTIONS:
Behavioral: Metacognitive Training (MCT) — The metacognitive group training program that will form the basis of the 16 session MCT intervention has been described in previous research (Moritz & Woodward 2007a; Moritz & Woodward 2007b; Moritz 2011) and can be obtained online at no cost (www.uke.de/mkt). This experimental intervention will consist of two 8-module cycles occurring twice a week for 8 weeks, for a total of 16 sessions. Each module will include a 45 to 60 minute instructor-led group session using PowerPoint slides and homework assignments to facilitate learning. Groups will consist of 4-10 subjects. Subjects will be able to attend the alternate (Cognitive Remediation) group after completion of the MCT group if they wish.
  Arms: Metacognitive Training for Psychosis
Behavioral: Cognitive Remediation (CR) — The CR group will use a computerized cognitive remediation program that has been used with schizophrenia patients, Scientific Brain Training Pro (SBT Pro; Vianin et al, 2010). Modules focus on attention, working memory, verbal memory, and planning and reasoning. Each session will incorporate psycho-educational group discussion of strategies, and individual work through exercises on personal tablet computers and personalized level of difficulty. The CR treatment will take place twice per week for 8 weeks, for a total of 16 sessions. Groups will consist of 4-10 subjects. Subjects will be able to attend MCT after completion of CR if they wish.
  Arms: Cognitive Remediation for Psychosis

SUMMARY:
Current Canadian Clinical Practice guidelines emphasize the need for effective psychosocial adjuncts to pharmacotherapy for schizophrenia (Canadian Psychiatric Association 2005). This randomized control trial seeks to contribute to the body of evidence supporting psychosocial treatments by assessing the effectiveness of metacognitive training (MCT) and cognitive remediation (CR) at treating the persistent positive and cognitive symptoms of schizophrenia. MCT is a therapy designed to improve patient awareness and insight into the cognitive biases that are frequently seen in schizophrenia; it has been associated with decreased psychopathology (specifically decreased positive symptoms) and improved psychosocial function. CR is a therapy designed to improve performance in a variety of neurocognitive functions such as attention, memory, and executive functioning; it has been associated with improved cognitive and psychosocial functioning. Both MCT and CR will be compared to treatment as usual (TAU) as done previously (Kumar er al., 2010; Moritz et al., 2011).

Hypotheses:

1. MCT will produce greater change in delusions (severity and conviction) than CR and TAU.
2. CR and MCT will produce greater change in social/everyday functioning than TAU.
3. CR will produce greater improvement in basic attention and memory measures relative to MCT and TAU.
4. MCT will produce greater reduction on tasks measuring targeted reasoning biases relative to CR and TAU.
5. CR will increase efficiency of functional networks on a working memory task relative to MCT and TAU.
6. MCT will lead to a greater decrease in the neural response to evidence matches relative to CR and TAU.

DETAILED DESCRIPTION:
Objectives:

The objectives of this research project is to assess the relative effectiveness of MCT and CR at treating the persistent positive symptoms of schizophrenia in a stable patient population. Specifically, we will use verified measures to examine the impact of these interventions on delusion conviction and severity, as well as on other features of interest, including insight and specific cognitive biases. We will use functional neuroimaging, both electroencephalography (EEG) and functional Magnetic Resonance Imaging (fMRI), to measure the changes in the neural responses while subjects are performing various cognitive tasks. It is expected that improvements in cognitive performance and function seen with MCT and CR correlate with select improvements in efficiency of particular brain networks. We anticipate a double dissociation, in that subjects with decreased positive symptoms following MCT may present with different patterns of activation than those with improved neurocognitive function following CR.

Procedures:

Recruitment will be done through inpatient and outpatient departments in Vancouver, British Columbia, Canada. Diagnosis of schizophrenia spectrum disorder will be confirmed using the MINI (Sheehan, 1998). Both inpatients and outpatients will be recruited; patients must be identified as suitable, as determined by their treating psychiatric team. This will suffice to obtain 50 subjects per condition over 5 years. Note that our intended sample size was originally 75 per group, which would allow for attrition and still give us an estimated 50 subjects with completed and valid behavioural and neuroimaging data.

Participants who complete the screening and baseline (pre-treatment) assessments will be randomly assigned to one of 3 conditions: 1) MCT, 2) CR, or 3) TAU. Randomization of subjects will occur as they complete their baseline assessments, and entry into the groups will involve a rolling intake model. Interventions will be administered twice weekly for 8 weeks. The groups will be run by Clinical Psychologists and PhD level psychology students. Allied health professionals, such as Occupational Therapists or Social Workers, may co-facilitate groups.

Baseline (pre-treatment), midpoint, and post-treatment assessments will include symptom and cognitive assessment, as well as self-reported measures, as outlined above. Patients who are willing and eligible will also be involved in three tasks in which we will record both fMRI data and EEG data.

fMRI scanning:

Participants will be prepared for EEG by trained graduate students, research staff, and fMRI technicians. Once in the scanner, the subject will perform three cognitive tasks which have been used extensively in previous research.

EEG recording:

Participants will be prepared for EEG by trained graduate students and research staff. The subjects will perform the same cognitive tasks as the fMRI procedure.

Measurements:

Symptom Ratings:

General psychopathology will be assessed using the Scale for the Assessment of Negative Symptoms (SANS; Andreasen, 1984) and the Scale for the Assessment of Positive Symptoms (SAPS; Andreasen, 1984). Delusion severity will be measured using the Delusions Scale of the Psychotic Symptom Rating Scales (PSYRATS; Haddock, McCarron, Tarrier, & Faragher, 1999). All symptom rating scales will be administered by trained raters blinded to the treatment allocations of subjects.

Self-Report Measures:

Patient depressive symptoms will be measured using the Beck Depression Inventory, Second Edition (BDI-II, Beck, 1996). Patient perception of their quality of life will be measured using the World Health Organisation Quality of Life scale (WHOQoL). Patient perception of stigma and its impact on their quality of life will be measured using the Internalized Stigma of Mental Illness scale (ISMI; Ritsher et al., 2003). Patient perceptions of self and self-esteem will be measured using the Rosenberg Self-Esteem Scale (RSES; Rosenberg, 1965).

Cognitive Biases

MCT for psychosis is fundamentally concerned with dysfunctional thinking in psychotic illnesses and it directly targets cognitive biases known to be involved in delusional thinking including the jumping to conclusions bias, the attributional bias, and the bias against disconfirmatory evidence. Two cognitive biases commonly seen in schizophrenia will be evaluated using the "jumping to conclusions (JTC) task" (also known as the "fisherman" task) and the "bias against disconfirmatory evidence (BADE)" task. These tasks were developed, in part, by the Principal Investigator and have been described in previous research (Lecomte & Woodward, 2005; Woodward 2006a; Woodward 2006b; Woodward 2007; Moritz & Woodward 2005; Woodward 2009).

The test of Premorbid Function (ToPF) is a word-reading task that will be used to estimate the premorbid intelligence (IQ) of the individual (Wechsler, 2011). The Wechsler Abbreviated Scale of Intelligence, Second Edition (WASI-II; Wechsler, 2011) will provide a measure of current intelligence (IQ). The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS; Randolph, 1998) will be used to review neurocognitive function of the individual, including attention, processing speed, working memory, verbal and visual memory. The trailmaking test will provide measures of basic attention, speed of processing, mental flexibility, and executive functioning (Reitan, 1992). The Controlled Oral Word Association test (COWAT; Benton et al., 1994) is a verbal fluency task that measures executive functioning.

Insight

The Beck Cognitive Insight Scale (BCIS; Beck, Baruch, Balter, Steer, & Warman, 2004) will be administered to evaluate patients' degree of insight into cognitive biases and limitations.

Functional Neuroimaging and Electroencephalography

Functional Magnetic Resonance Imaging (fMRI) and Electroencephalography (EEG) will be used to assess the relative involvement and activation of different neural networks. The Sternberg Working Memory Task will be used in order to quantify the level of efficiency of the neural networks responsible for working memory (Metzak et al., 2012). Two Evidence Matching Tasks (e.g., the "fish task" and the "bias against discomfirmatory evidence (BADE) task") will be used in order to quantify the reactivity of the neural networks responsible for evidence matching (e.g., anterior-cingulate-based network; Woodward et al., 2008).

Feedback from Participants

After the final session in active treatment conditions, patients will be asked to complete a questionnaire comprising 10 questions on acceptance and subjective efficacy (Moritz & Woodward 2007a). Data accumulated therein will be used together with frequency of unattended sessions to establish acceptability and feasibility of the various treatment conditions.

Statistical Analysis

Rolling group intake and facilitation will allow for two to four, two-month cycles of each condition per year for 5 years, which should allow us to obtain 75 subjects per condition. This would allow for possible attrition, and still give us an estimated 50 subjects per condition (MCT, CR, TAU), which is sufficient to produce a power of 0.8 to detect a large effect in a three group means comparison design (Cohen 1992) using p=0.05 as the cutoff for significance.

Notes on Actual Enrollment (As the Study Has Been Terminated)

Out of the intended enrollment of 225 subjects (75 subjects per group), 129 subjects were actually enrolled. Of these 129 subjects actually enrolled, approximately 60 subjects have a completed dataset.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 19 to 60 years
2. Diagnosis of schizophrenia, schizoaffective disorder or schizophreniform disorder.
3. Diagnosis of mood disorder with current psychosis.

Exclusion Criteria:

1. An inability to read and write in English. Participants must be have used English on a daily basis for at least 5 years, and must be able to understand the consent form and give written consent.
2. A history of severe neurological disorder and those with severe manifestations of hostility, megalomania, formal thought disorder and suspiciousness.
3. Subjects who are obtaining ongoing electroconvulsive therapy (ECT)
4. Subjects who are consistently disrupting the rest of the group might be asked to leave, this will be at the discretion of the group instructor.

In addition to the group exclusion criteria, the exclusion criteria for Neuroimaging (fMRI):

1. History of brain damage or other medical problems that may affect comprehension (e.g., seizure disorders, stroke, aneurysm, brain tumor, etc.)
2. Psychosis that is a direct consequence of substance abuse.
3. Currently suffer from severe substance dependence.
4. Surgery within the last 6 weeks.
5. Surgery to the brain, heart or eyes.
6. Metal implants
7. Metal fragments in or near your eyes.
8. Pregnant.
9. Recent serious concussion, or loss of consciousness of more than 10 minutes.
10. Colour blind

In addition to the group exclusion criteria, the exclusion criteria for Neuroimaging EEG:

1. History of brain damage or other medical problems that may affect comprehension (e.g., seizure disorders, stroke, aneurysm, brain tumor, etc.)
2. Recent serious concussion, or loss of consciousness of more than 10 minutes
3. Currently suffer from severe substance dependence.
4. Colour blind

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Delusion Severity | 8-12 weeks (post-treatment) relative to baseline (pre-treatment)
  Delusion severity will be measured using the Delusions Scale of the Psychotic Symptom Rating Scales (PSYRATS; Haddock, McCarron, Tarrier, & Faragher, 1999). The PSYRATS Delusion Scale measures more specific aspects of delusions such as conviction and impact on thinking.

SECONDARY OUTCOMES:
Symptom Ratings | 4 weeks (midpoint of therapy) relative to baseline (pre-treatment)
  General psychopathology will be assessed using the Scale for the Assessment of Negative Symptoms (SANS; Andreasen, 1984) and the Scale for the Assessment of Positive Symptoms (SAPS; Andreasen, 1984). Patient depressive symptoms will be measured using the Beck Depression Inventory, Second Edition (BDI-II; Beck, 1996). Patient perception of their quality of life will be measured using the World Health Organisation Quality of Life Scale (WHOQoL). Patient perception of stigma and its impact on their quality of life will be measured using the Internalized Stigma of Mental Illness scale (Ritsher et al, 2003). All symptom ratings will be administered by trained raters blinded to the treatment allocation of subjects.
Symptom Ratings | 8-12 weeks (post-treatment) relative to baseline (pre-treatment)
  General psychopathology will be assessed using the Scale for the Assessment of Negative Symptoms (SANS; Andreasen, 1984) and the Scale for the Assessment of Positive Symptoms (SAPS; Andreasen, 1984). Patient depressive symptoms will be measured using the Beck Depression Inventory, Second Edition (BDI-II, Beck 1996). Patient perception of their quality of life will be measured using the World Health Organization Quality of Life scale (WHOQoL). Patient perception of stigma and its impact on their quality of life will be measured using the Internalized Stigma of Mental Illness scale (Ritsher et al, 2003). All symptom rating scales will be administered by trained raters blinded to the treatment allocation of subjects.
Cognitive Function | Pre-treatment (prior to commencement of therapy)
  The Test of Premorbid Function (ToPF) is a word-reading task that will be used to estimate the premorbid intelligence (IQ) of the individual (Wechsler, 2011). The Wechsler Abbreviated Scale of Intelligence, Second Edition (WASI-II; Wechsler, 2011) will provide a measure of current cognitive function (or intelligence). The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS; Randolph, 1998) will be used to review neurocognitive function of the individual, including attention, processing speed, working memory, verbal and visual memory. Trailmaking Test will provide measures of basic attention, speed of processing, mental flexibility, and executive functioning. The Controlled Oral Word Association test (COWAT) is a verbal fluency task that measures executive functioning. The Letter Number Sequencing test measures working memory, with ability to recall and organize a sequence of letters and numbers (Wechsler, 2011).
Cognitive Function | 4 weeks (midpoint of therapy) relative to baseline (pre-treatment)
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS; Randolph, 1998) will be used to review neurocognitive function of the individual, including attention, processing speed, working memory, verbal and visual memory. Trailmaking Test will provide measures of basic attention, speed of processing, mental flexibility, and executive functioning. The Controlled Oral Word Association test (COWAT) is a verbal fluency task that measures executive functioning.
Cognitive Function | 8-12 weeks (post-treatment) relative to baseline (pre-treatment)
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS; Randolph, 1998) will be used to review neurocognitive function of the individual, including attention, processing speed, working memory, verbal and visual memory. Trailmaking Test will provide measures of basic attention, speed of processing, mental flexibility, and executive functioning. The Controlled Oral Word Association test (COWAT) is a verbal fluency task that measures executive functioning. The Letter Number Sequencing test is a measure of working memory, with the ability to recall and organize a sequence of letters and numbers (Wechsler, 2011).
Cognitive Bias | 4 weeks (midpoint of therapy) relative to baseline (pre-treatment)
  Two cognitive biases commonly seen in schizophrenia will be evaluated using the "jumping to conclusions (JTC)" tasks and the "bias against disconfirmatory evidence (BADE)" tasks. These tasks were developed, in part, by the principal investigator and have been described in previous research (Lecomte & Woodward 2005; Woodward 2006a; Woodward 2006b; Woodward 2007; Moritz & Woodward 2005; Woodward 2009).
Cognitive Bias | 8-12 weeks (post-treatment) relative to baseline (pre-treatment)
  Two cognitive biases commonly seen in schizophrenia will be evaluated using the "jumping to conclusions (JTC) scale" and the "bias against disconfirmatory evidence (BADE)" tasks. These tasks were developed, in part, by the principal investigator and have been described in previous research (Lecomte & Woodward 2005; Woodward 2006a; Woodward 2006b; Woodward 2007; Moritz & Woodward 2005; Woodward 2009).
Insight | 4 weeks (midpoint of therapy) relative to baseline (pre-treatment)
  The Beck Cognitive Insight Scale (BCIS; Beck, Baruch, Balter, Steer, & Warman 2004) will be administered to evaluate patients' degree of insight into cognitive biases and limitations.
Insight | 8-12 weeks (post-treatment) relative to baseline (pre-treatment)
  The Beck Cognitive Insight Scale (BCIS; Beck, Baruch, Balter, Steer, & Warman 2004) will be administered to evaluate patients' degree of insight into cognitive biases and limitations.
Psychosocial/Everyday Functioning | 4 weeks (midpoint of therapy) relative to baseline (pre-treatment)
  Subjects social functioning in daily interactions will be assessed using the Social Functioning Scale (SFS; Birchwood et al., 1990).
Psychosocial/Everyday Functioning | 8-12 weeks (post-treatment) relative to baseline (pre-treatment)
  Subjects social functioning in daily interactions will be assessed using the Social Functioning Scale (SFS; Birchwood et al., 1990).
Feasibility and acceptability | 8-12 weeks (post-treatment)
  After the final session in active treatment conditions, patients will be asked to complete a questionnaire comprising 10 questions on acceptance and subjective efficacy (Moritz & Woodward, 2007a). Data accumulated therein will be used together with frequency of unattended sessions to establish acceptability and feasibility of the various treatment conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Woodward, PhD, Principal Investigator — University of British Columbia; Mahesh Menon, PhD, RPsych, Principal Investigator — University of British Columbia
Locations (1):
- UBC Hospital - Detwiller Pavilion, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Barrowclough C, Haddock G, Lobban F, Jones S, Siddle R, Roberts C, Gregg L. Group cognitive-behavioural therapy for schizophrenia. Randomised controlled trial. Br J Psychiatry. 2006 Dec;189:527-32. doi: 10.1192/bjp.bp.106.021386. PMID 17139037
- [Background] Beck AT, Baruch E, Balter JM, Steer RA, Warman DM. A new instrument for measuring insight: the Beck Cognitive Insight Scale. Schizophr Res. 2004 Jun 1;68(2-3):319-29. doi: 10.1016/S0920-9964(03)00189-0. PMID 15099613
- [Background] Bechdolf A, Knost B, Nelson B, Schneider N, Veith V, Yung AR, Pukrop R. Randomized comparison of group cognitive behaviour therapy and group psychoeducation in acute patients with schizophrenia: effects on subjective quality of life. Aust N Z J Psychiatry. 2010 Feb;44(2):144-50. doi: 10.3109/00048670903393571. PMID 20113303
- [Background] Cohen J. A power primer. Psychol Bull. 1992 Jul;112(1):155-9. doi: 10.1037//0033-2909.112.1.155. PMID 19565683
- [Background] Haddock G, McCarron J, Tarrier N, Faragher EB. Scales to measure dimensions of hallucinations and delusions: the psychotic symptom rating scales (PSYRATS). Psychol Med. 1999 Jul;29(4):879-89. doi: 10.1017/s0033291799008661. PMID 10473315
- [Background] Lecomte T, Leclerc C, Corbiere M, Wykes T, Wallace CJ, Spidel A. Group cognitive behavior therapy or social skills training for individuals with a recent onset of psychosis? Results of a randomized controlled trial. J Nerv Ment Dis. 2008 Dec;196(12):866-75. doi: 10.1097/NMD.0b013e31818ee231. PMID 19077853
- [Background] Liddle PF, Ngan ET, Duffield G, Kho K, Warren AJ. Signs and Symptoms of Psychotic Illness (SSPI): a rating scale. Br J Psychiatry. 2002 Jan;180:45-50. doi: 10.1192/bjp.180.1.45. PMID 11772851
- [Background] Moritz S, Woodward TS. Jumping to conclusions in delusional and non-delusional schizophrenic patients. Br J Clin Psychol. 2005 Jun;44(Pt 2):193-207. doi: 10.1348/014466505X35678. PMID 16004654
- [Background] Moritz S, Woodward TS. Metacognitive training in schizophrenia: from basic research to knowledge translation and intervention. Curr Opin Psychiatry. 2007 Nov;20(6):619-25. doi: 10.1097/YCO.0b013e3282f0b8ed. PMID 17921766
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Tarrier N, Yusupoff L, Kinney C, McCarthy E, Gledhill A, Haddock G, Morris J. Randomised controlled trial of intensive cognitive behaviour therapy for patients with chronic schizophrenia. BMJ. 1998 Aug 1;317(7154):303-7. doi: 10.1136/bmj.317.7154.303. PMID 9685273
- [Background] Woodward TS, Moritz S, Chen EY. The contribution of a cognitive bias against disconfirmatory evidence (BADE) to delusions: a study in an Asian sample with first episode schizophrenia spectrum disorders. Schizophr Res. 2006 Apr;83(2-3):297-8. doi: 10.1016/j.schres.2006.01.015. Epub 2006 Mar 2. No abstract available. PMID 16513331
- [Background] Woodward TS, Moritz S, Cuttler C, Whitman JC. The contribution of a cognitive bias against disconfirmatory evidence (BADE) to delusions in schizophrenia. J Clin Exp Neuropsychol. 2006 May;28(4):605-17. doi: 10.1080/13803390590949511. PMID 16624787
- [Background] Woodward TS, Buchy L, Moritz S, Liotti M. A bias against disconfirmatory evidence is associated with delusion proneness in a nonclinical sample. Schizophr Bull. 2007 Jul;33(4):1023-8. doi: 10.1093/schbul/sbm013. Epub 2007 Mar 8. PMID 17347526
- [Background] Woodward TS, Munz M, LeClerc C, Lecomte T. Change in delusions is associated with change in "jumping to conclusions". Psychiatry Res. 2009 Dec 30;170(2-3):124-7. doi: 10.1016/j.psychres.2008.10.020. Epub 2009 Nov 10. PMID 19906443
- [Background] Wykes T, Parr AM, Landau S. Group treatment of auditory hallucinations. Exploratory study of effectiveness. Br J Psychiatry. 1999 Aug;175:180-5. doi: 10.1192/bjp.175.2.180. PMID 10627803
- [Background] Canadian Psychiatric Association. Clinical practice guidelines. Treatment of schizophrenia. Can J Psychiatry. 2005 Nov;50(13 Suppl 1):7S-57S. No abstract available. PMID 16529334
- [Background] Lecomte, T., Woodward, T. S., & Leclerc, C. (2005). Changes in the jumping-to-conclusions bias are associated with changes in delusions: A longitudinal study involving cognitive behavioural therapy [abstract]. Schizophrenia Research, 31, 365.
- [Background] Moritz, S., & Woodward, T. S. (2007a). Metacognitive training for schizophrenia patients (MCT): A pilot study on feasibility, treatment adherence, and subjective efficacy. German Journal of Psychiatry, 10, 69-78.
- [Background] Moritz S, Veckenstedt R, Randjbar S, Vitzthum F, Woodward TS. Antipsychotic treatment beyond antipsychotics: metacognitive intervention for schizophrenia patients improves delusional symptoms. Psychol Med. 2011 Sep;41(9):1823-32. doi: 10.1017/S0033291710002618. Epub 2011 Jan 28. PMID 21275083
- [Background] Bartholomeusz CF, Allott K. Neurocognitive and social cognitive approaches for improving functional outcome in early psychosis: theoretical considerations and current state of evidence. Schizophr Res Treatment. 2012;2012:815315. doi: 10.1155/2012/815315. Epub 2012 Apr 5. PMID 22966447
- [Background] Wykes T, Huddy V, Cellard C, McGurk SR, Czobor P. A meta-analysis of cognitive remediation for schizophrenia: methodology and effect sizes. Am J Psychiatry. 2011 May;168(5):472-85. doi: 10.1176/appi.ajp.2010.10060855. Epub 2011 Mar 15. PMID 21406461
- [Background] McGurk SR, Twamley EW, Sitzer DI, McHugo GJ, Mueser KT. A meta-analysis of cognitive remediation in schizophrenia. Am J Psychiatry. 2007 Dec;164(12):1791-802. doi: 10.1176/appi.ajp.2007.07060906. PMID 18056233